CLINICAL TRIAL: NCT00807833
Title: Cerebral Blood Flow (CBF) Disturbances Following Traumatic Brain Injury (TBI) and Subarachnoid Hemorrhage (SAH)
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Dott. Giuseppe Citerio, MD, Azienda Ospedaliera San Gerardo di Monza
Other Study IDs: 08-007
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
Keywords: SAH; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CBF measurement: It is a "proof of concept" study, aimed to evaluate whether the "optimal CPP", defined by the best PRx, corresponds to the acceptable CBF values.
  Patients admitted with the diagnosis of TBI and SAH in for whom ICP and CPP needs to be monitored on clinical ground will be also monitored with a TD probe and routinely tested for cerebral autoregulation, thus obtaining the CBF corresponding at a given the "best CPP" and autoregulation status.

SUMMARY:
It is a "proof of concept" study, aimed to evaluate whether the "optimal CPP", defined by the best PRx, corresponds to the acceptable CBF values in patients affected by CBF disfunction caused by TBI or SAH.

DETAILED DESCRIPTION:
Cerebral blood flow (CBF) disturbances are common following TBI and SAH. The occurrence of CBF derangements is detrimental for the neurological outcome in both settings, but the management of neurologically critically ill patients does not involve CBF measure routinely. Cerebrovascular autoregulation, can be assessed by the cerebrovascular pressure-reactivity index (PRx) that point out the response of ICP to spontaneous changes in arterial blood pressure (ABP). Autoregulation has been proven to be a powerful protective mechanism. Adding together the information on CBF and autoregulation, might drive clinical strategy in exceptionally noteworthy and innovative way. Currently, a novel Thermal Diffusion (TDP) microprobe has been introduced for the continuous bedside monitoring of regional CBF: TDP is a promising technique in the reliable detection of flow derangements at the patient's bedside.

It is a "proof of concept" study, aimed to evaluate whether the "optimal CPP", defined by the best PRx, corresponds to the acceptable CBF values.

Patients admitted with the diagnosis of TBI and SAH in for whom ICP and CPP needs to be monitored on clinical ground will be also monitored with a TD probe and routinely tested for cerebral autoregulation, thus obtaining the CBF corresponding at a given the "best CPP" and autoregulation status.

Continuous CBF measures and PRx monitoring may allow more accurate identification and early detection of adverse cerebral conditions. This approach may bring us a step closer to the goal of outcome improvements in patients suffering from intracranial insult.

ELIGIBILITY:
Inclusion criteria:

* Patients admitted with the diagnosis of SAH and requiring intensive monitoring, and ICP probe.
* Patients admitted diagnosis of severe TBI and requiring intensive monitoring, and ICP probe.

Exclusion criteria:

* Age < 16 years
* Previous SAH, brain surgery, stroke, brain trauma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with the diagnosis of TBI and SAH in for whom ICP and CPP needs to be monitored on clinical ground will be also monitored with a TD probe and routinely tested for cerebral autoregulation, thus obtaining the CBF corresponding at a given the "best CPP" and autoregulation status. Continuous CBF measures and PRx monitoring may allow more accurate identification and early detection of adverse cerebral conditions. This approach may bring us a step closer to the goal of outcome improvements in patients suffering from intracranial insult.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the "optimal CPP", defined by PRx, corresponds to the acceptable CBF values | one week

SECONDARY OUTCOMES:
Compare in cohort group PRx/CPP curve to CBFx/CPP curve.The "CBFx" index is defined as the moving correlation between slow waves in CPP and CBF | one week

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, DM, Principal Investigator — Azienda Ospedaliera San Gerardo Monza
Locations (1):
- Azienda Ospedaliera San Gerardo, Monza, Italy, Italy

REFERENCES:
- [Background] Claassen J, Vu A, Kreiter KT, Kowalski RG, Du EY, Ostapkovich N, Fitzsimmons BF, Connolly ES, Mayer SA. Effect of acute physiologic derangements on outcome after subarachnoid hemorrhage. Crit Care Med. 2004 Mar;32(3):832-8. doi: 10.1097/01.ccm.0000114830.48833.8a. PMID 15090970
- [Background] Vespa P, Bergsneider M, Hattori N, Wu HM, Huang SC, Martin NA, Glenn TC, McArthur DL, Hovda DA. Metabolic crisis without brain ischemia is common after traumatic brain injury: a combined microdialysis and positron emission tomography study. J Cereb Blood Flow Metab. 2005 Jun;25(6):763-74. doi: 10.1038/sj.jcbfm.9600073. PMID 15716852
- [Background] Coles JP, Fryer TD, Smielewski P, Chatfield DA, Steiner LA, Johnston AJ, Downey SP, Williams GB, Aigbirhio F, Hutchinson PJ, Rice K, Carpenter TA, Clark JC, Pickard JD, Menon DK. Incidence and mechanisms of cerebral ischemia in early clinical head injury. J Cereb Blood Flow Metab. 2004 Feb;24(2):202-11. doi: 10.1097/01.WCB.0000103022.98348.24. PMID 14747747
- [Background] Czosnyka M, Pickard JD. Monitoring and interpretation of intracranial pressure. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):813-21. doi: 10.1136/jnnp.2003.033126. PMID 15145991
- [Background] Lam JM, Smielewski P, Czosnyka M, Pickard JD, Kirkpatrick PJ. Predicting delayed ischemic deficits after aneurysmal subarachnoid hemorrhage using a transient hyperemic response test of cerebral autoregulation. Neurosurgery. 2000 Oct;47(4):819-25; discussions 825-6. doi: 10.1097/00006123-200010000-00004. PMID 11014420
- [Background] Hutchinson PJ, Al-Rawi PG, O'Connell MT, Gupta AK, Maskell LB, Hutchinson DB, Pickard JD, Kirkpatrick PJ. Monitoring of brain metabolism during aneurysm surgery using microdialysis and brain multiparameter sensors. Neurol Res. 1999 Jun;21(4):352-8. doi: 10.1080/01616412.1999.11740943. PMID 10406006
- [Background] Weyer GW, Nolan CP, Macdonald RL. Evidence-based cerebral vasospasm management. Neurosurg Focus. 2006 Sep 15;21(3):E8. doi: 10.3171/foc.2006.21.3.8. PMID 17029347
- [Background] Longstreth WT Jr, Nelson LM, Koepsell TD, van Belle G. Clinical course of spontaneous subarachnoid hemorrhage: a population-based study in King County, Washington. Neurology. 1993 Apr;43(4):712-8. doi: 10.1212/wnl.43.4.712. PMID 8469328
- [Background] Biller J, Toffol GJ, Kassell NF, Adams HP Jr, Beck DW, Boarini DJ. Spontaneous subarachnoid hemorrhage in young adults. Neurosurgery. 1987 Nov;21(5):664-7. doi: 10.1227/00006123-198711000-00011. PMID 3696399
- [Background] Linn FH, Rinkel GJ, Algra A, van Gijn J. Incidence of subarachnoid hemorrhage: role of region, year, and rate of computed tomography: a meta-analysis. Stroke. 1996 Apr;27(4):625-9. doi: 10.1161/01.str.27.4.625. PMID 8614919
- [Background] Robertson CS. Management of cerebral perfusion pressure after traumatic brain injury. Anesthesiology. 2001 Dec;95(6):1513-7. doi: 10.1097/00000542-200112000-00034. No abstract available. PMID 11748413
- [Background] Howells T, Elf K, Jones PA, Ronne-Engstrom E, Piper I, Nilsson P, Andrews P, Enblad P. Pressure reactivity as a guide in the treatment of cerebral perfusion pressure in patients with brain trauma. J Neurosurg. 2005 Feb;102(2):311-7. doi: 10.3171/jns.2005.102.2.0311. PMID 15739560
- [Background] Soehle M, Jaeger M, Meixensberger J. Online assessment of brain tissue oxygen autoregulation in traumatic brain injury and subarachnoid hemorrhage. Neurol Res. 2003 Jun;25(4):411-7. doi: 10.1179/016164103101201580. PMID 12870270
- [Background] Jaeger M, Schuhmann MU, Soehle M, Nagel C, Meixensberger J. Continuous monitoring of cerebrovascular autoregulation after subarachnoid hemorrhage by brain tissue oxygen pressure reactivity and its relation to delayed cerebral infarction. Stroke. 2007 Mar;38(3):981-6. doi: 10.1161/01.STR.0000257964.65743.99. Epub 2007 Feb 1. PMID 17272764
- [Background] Vajkoczy P, Horn P, Thome C, Munch E, Schmiedek P. Regional cerebral blood flow monitoring in the diagnosis of delayed ischemia following aneurysmal subarachnoid hemorrhage. J Neurosurg. 2003 Jun;98(6):1227-34. doi: 10.3171/jns.2003.98.6.1227. PMID 12816269
- [Background] Vajkoczy P, Roth H, Horn P, Lucke T, Thome C, Hubner U, Martin GT, Zappletal C, Klar E, Schilling L, Schmiedek P. Continuous monitoring of regional cerebral blood flow: experimental and clinical validation of a novel thermal diffusion microprobe. J Neurosurg. 2000 Aug;93(2):265-74. doi: 10.3171/jns.2000.93.2.0265. PMID 10930012
- [Background] Vajkoczy P, Horn P, Bauhuf C, Munch E, Hubner U, Ing D, Thome C, Poeckler-Schoeninger C, Roth H, Schmiedek P. Effect of intra-arterial papaverine on regional cerebral blood flow in hemodynamically relevant cerebral vasospasm. Stroke. 2001 Feb;32(2):498-505. doi: 10.1161/01.str.32.2.498. PMID 11157189
- [Background] Thome C, Vajkoczy P, Horn P, Bauhuf C, Hubner U, Schmiedek P. Continuous monitoring of regional cerebral blood flow during temporary arterial occlusion in aneurysm surgery. J Neurosurg. 2001 Sep;95(3):402-11. doi: 10.3171/jns.2001.95.3.0402. PMID 11565860